CLINICAL TRIAL: NCT02687802
Title: Respiratory Mechanics and Patient-ventilator Asynchrony Index in Patients With Invasive Mechanical Ventilation
Acronym: EpiSync
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015/19122-4
Record Dates: First submitted 2016-01-18; First posted 2016-02-22 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Insufficiency
Keywords: respiratory mechanics; Respiratory Insufficiency; artificial, ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanical ventilation: Patients under mechanical ventilation for more than 24h
  Interventions: Other: mechanical ventilation

INTERVENTIONS:
Other: mechanical ventilation — we will measure static resistance, compliance and intrinsic positive end-expiratory pressure (PEEP) and other variables as risk factors for asynchrony occurrence

SUMMARY:
The objective of the study is to estimate the incidence of asynchrony and to assess its relationship with respiratory mechanics. This will be a prospective cohort study, including patients under invasive mechanical ventilation. Within 48h post intubation, the investigators will record the values of intrinsic positive end-expiratory pressure, pulmonary compliance and resistance. Participants will be followed up from intubation to mechanical ventilation liberation. The investigators will register clinical signs of asynchrony and record ventilator waveforms continuously and quantify patient-ventilator asynchrony. The investigators will calculate the total asynchrony index (AI) and of each asynchrony type (ineffective triggering, double triggering, auto triggering, short cycling and prolonged cycling). Participants will be followed up until hospital discharge.

DETAILED DESCRIPTION:
Patient-ventilator asynchrony is common in patients under invasive mechanical ventilation, present between 10 and 80% of all respiratory cycles, and is associated with adverse clinical outcomes, such as delay in the weaning process, increased complications of mechanical ventilation, with possible impact on survival. The objective of this study is to estimate the incidence of asynchrony and to assess its relationship with respiratory mechanics. This will be a prospective cohort study, including all patients under invasive mechanical ventilation admitted at Respiratory ICU at Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo (USP), during the study period. Within 48h post intubation, the investigators will record the values of intrinsic positive end-expiratory pressure, pulmonary compliance and resistance. Participants will be followed up from intubation to mechanical ventilation liberation. The investigators will register clinical signs of asynchrony and record ventilator waveforms continuously. The ventilator waveforms will be captured directly from ventilator and processed by dedicated software, without direct contact with patients. Later, ventilator waveforms will be analyzed to quantify patient-ventilator asynchrony. The investigators will calculate the total asynchrony index (AI) and of each asynchrony type (ineffective triggering, double triggering, auto triggering, short cycling and prolonged cycling). Participants will be followed up until hospital discharge, and the investigators will record duration of mechanical ventilation, the use of non-invasive ventilation post-extubation, reintubation, tracheostomy, ICU and hospital length of stay and survival. With this project, the investigators will estimate the incidence and magnitude of patient-ventilator asynchrony and its association with clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Recent mechanical ventilation (less than 72 hours)
* Expectation of mechanical ventilation for more than 24 hours
* Age ≥ 18 years old

Exclusion Criteria:

* High flow Bronchopleural fistula
* Thoracic or abdominal deformities that could compromise the accuracy of respiratory mechanics measurement
* Impossibility to measure respiratory mechanics
* Tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients intubated and under invasive mechanical ventilation in a University hospital ICU
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
asynchrony index | from study inclusion until the date of extubation or date of death from any cause, whichever comes first, up to 28 days
  asynchrony index will be calculated as the number of major asynchrony events divided by total number of respiratory cycles

SECONDARY OUTCOMES:
Clinical signs of patient-ventilator asynchrony | daily, from study inclusion until the date of extubation or date of death from any cause, whichever comes first, up to 28 days
  a standardized questionnaire will be used to evaluate the presence of clinically significant patient-ventilator asynchrony. Trained investigators will observe participant´s breathing pattern and other clinical signs of patient-ventilator asynchrony and score each item as absent (0) or present (1). Then, they will visual inspection of ventilator waveforms on the ventilator screen for a 5 minute observation period, looking for missed efforts, double triggering, auto-triggering, cycling delay and premature cycling, as previously defined. If they observe more than 1 asynchrony event for every 10 respiratory cycles, they will rate this item as present (1), otherwise, they will rate it as absent (0).
ventilation free-days | 28 days
  number of days alive and off the ventilator up to day 28
tracheostomy rate | up to 90 days
  performance of surgical or bronchoscopy-guided tracheotomy
Survival rate | at 28 and 90 days
  survival from intubation up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Ferreira, MD, Principal Investigator — Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Hospital das Clínicas -HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No individual personal data will be disclosed

REFERENCES:
- [Derived] Sousa MLA, Magrans R, Hayashi FK, Blanch L, Kacmarek RM, Ferreira JC. Predictors of asynchronies during assisted ventilation and its impact on clinical outcomes: The EPISYNC cohort study. J Crit Care. 2020 Jun;57:30-35. doi: 10.1016/j.jcrc.2020.01.023. Epub 2020 Jan 21. PMID 32032901
- [Derived] Sousa MLA, Magrans R, Hayashi FK, Blanch L, Kacmarek RM, Ferreira JC. EPISYNC study: predictors of patient-ventilator asynchrony in a prospective cohort of patients under invasive mechanical ventilation - study protocol. BMJ Open. 2019 May 22;9(5):e028601. doi: 10.1136/bmjopen-2018-028601. PMID 31123002